CLINICAL TRIAL: NCT03195881
Title: Post Cardiac Arrest Neuroprognostication Using the Diameter of Optic Nerve Sheath Via Ocular ultRAsound
Brief Title: Neuroprognostication Using Optic Nerve Sheath Diameter
Acronym: PANDORA
Status: Completed | Type: Observational
Sponsor: TriHealth Inc. (Other)
Collaborators: TriHealth Hatton Research Institute (Other); Jocelyn LaMar (Unknown); Emily Craver (Unknown)
Responsible Party: Sponsor
Other Study IDs: 16-057
Record Dates: First submitted 2017-06-02; First posted 2017-06-22 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2019-08

CONDITIONS: Heart Arrest; Intracranial Pressure Increase
MeSH Terms: conditions — Heart Arrest; Intracranial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ocular ultrasound — Post-cardiopulmonary arrest patients meeting inclusion/exclusion criteria for targeted temperature management will undergo ocular ultrasound at three time points: within 6 hours (h) of initiation of hypothermic protocol, between 10-24 h after hypothermic protocol initiation, and between 24-36 h after hypothermic protocol initiation.

SUMMARY:
This study investigates the relationship between optic nerve sheath diameter and increased intracranial pressure and its effect on neurologic outcome in post-cardiopulmonary arrest patients.

DETAILED DESCRIPTION:
This study involves patients who have experienced either an in-hospital or out-of-hospital cardiopulmonary arrest, and who meet the 2015 American Heart Association (AHA) inclusion/exclusion criteria for targeted temperature management [i.e., they are comatose or exhibit no meaningful response to verbal commands with return of spontaneous circulation (ROSC) after cardiac arrest]. After induction of hypothermia protocol after cardiopulmonary arrest (i.e., targeted temperature management), patients will undergo ocular ultrasound at three time points.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years of age
* Patient has experienced either an in-hospital or out-of-hospital cardiopulmonary arrest
* Patient is comatose or exhibits lack of meaningful response to verbal commands with return of spontaneous circulation (ROSC) after cardiopulmonary arrest
* Patient must meet all inclusion criteria as deemed by physician and the 2015 American Heart Association standards for targeted temperature management (TTM) following cardiopulmonary arrest

Exclusion Criteria:

* Patient < 18 years of age
* Patient does not meet inclusion criteria for targeted temperature management (TTM)
* Unable to obtain consent from Legal Authorized Representative (LAR)
* Patient has a Do Not Resuscitate (DNR) order or a Do Not Intubate (DNI) order at the time of consent
* Patient has uncontrollable bleeding
* Patient is able to follow verbal commands
* Patient has another medical condition creating increased ocular pressure, as deemed by physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female post-cardiopulmonary arrest patients ≥ 18 years of age
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
Optic nerve sheath diameter | 0-6 hours after hypothermic protocol initiation
  Optic nerve sheath diameter within 6 hours of hypothermic protocol initiation

SECONDARY OUTCOMES:
Optic nerve sheath diameter | 10-24 hours after hypothermic protocol initiation
  Optic nerve sheath diameter 10-24 hours after hypothermic protocol initiation
Optic nerve sheath diameter | 24-36 hours after hypothermic protocol initiation
  Optic nerve sheath diameter 24-36 hours after hypothermic protocol initiation

OTHER OUTCOMES:
Modified Rankin Scale | Through day 2
  Measure of degree of disability or dependence in daily activities on day of informed consent
Modified Rankin Scale | Through 6 weeks
  Measure of degree of disability or dependence in daily activities on day of discharge from ICU'
Modified Rankin Scale | Up to 26 weeks
  Measure of degree of disability or dependence in daily activities six months after discharge from ICU
Cerebral Performance Category | Through day 2
  Measure of neurologic outcome following cardiac arrest on day of informed consent
Cerebral Performance Category | Through 6 weeks
  Measure of neurologic outcome following cardiac arrest on day of discharge from ICU
Cerebral Performance Category | Up to 26 weeks
  Measure of neurologic outcome following cardiac arrest six months after discharge from ICU

CONTACTS AND LOCATIONS:
Overall Officials: Lori Reid, MSN RN CCRC, Study Director — TriHealth Hatton Research Institute
Locations (1):
- Bethesda North TriHealth Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moretti R, Pizzi B. Ultrasonography of the optic nerve in neurocritically ill patients. Acta Anaesthesiol Scand. 2011 Jul;55(6):644-52. doi: 10.1111/j.1399-6576.2011.02432.x. Epub 2011 Apr 4. PMID 21463263
- [Background] Perkes I, Baguley IJ, Nott MT, Menon DK. A review of paroxysmal sympathetic hyperactivity after acquired brain injury. Ann Neurol. 2010 Aug;68(2):126-35. doi: 10.1002/ana.22066. PMID 20695005
- [Background] Rittenberger JC, Raina K, Holm MB, Kim YJ, Callaway CW. Association between Cerebral Performance Category, Modified Rankin Scale, and discharge disposition after cardiac arrest. Resuscitation. 2011 Aug;82(8):1036-40. doi: 10.1016/j.resuscitation.2011.03.034. Epub 2011 Apr 13. PMID 21524837
- [Background] Taccone F, Cronberg T, Friberg H, Greer D, Horn J, Oddo M, Scolletta S, Vincent JL. How to assess prognosis after cardiac arrest and therapeutic hypothermia. Crit Care. 2014 Jan 14;18(1):202. doi: 10.1186/cc13696. PMID 24417885
- [Background] Wang LJ, Yao Y, Feng LS, Wang YZ, Zheng NN, Feng JC, Xing YQ. Noninvasive and quantitative intracranial pressure estimation using ultrasonographic measurement of optic nerve sheath diameter. Sci Rep. 2017 Feb 7;7:42063. doi: 10.1038/srep42063. PMID 28169341